CLINICAL TRIAL: NCT00232687
Title: A Comparative, Randomized, Open-Label, Multicenter Study on the Efficacy and Safety of Switch Treatment With Aripiprazole in Schizophrenic Out-patients Who Are Experiencing Insufficient Efficacy With Risperidone and/or Safety and Tolerability Issues, While on Risperidone
Brief Title: A Switch Study of BMS-337039 in Schizophrenic Out-patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN138-169
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2012-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

ARMS (2):
- A1 (Active Comparator)
  Interventions: Drug: Aripiprazole
- A2 (Active Comparator)
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Tablets, Oral, 15 mg fixed dose (week 1-5) flexible dose 10-30 mg (week 6-12), once daily, 12 weeks.
  Other Names: Abilify
  Arms: A1
Drug: Aripiprazole — Tablets, Oral, Uptitration: 5 mg (week 1), 10 mg (week 2 and 3), 15 mg(week 4 and 5) flexible 10-30mg from week 6-12, once daily, 12 weeks.
  Other Names: Abilify
  Arms: A2

SUMMARY:
The purpose of this clinical research study is to evaluate the safety and tolerability of two switching strategies from risperidone to aripiprazole over a period of 12 weeks in out-patients who are treated in a general psychiatric practice setting and who are currently experiencing efficacy and/or safety/tolerability issues while on risperidone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of schizophrenia as defined by DSM-IV-TR2 criteria
* Out-patients who have been taking Risperidone for minimum 6 weeks who are not optimally controlled and/or experiencing safety/tolerability issues with Risperidone
* Men and women, aged 18 - 65 years

Exclusion Criteria:

* Patients who are at risk for committing suicide
* Patients with a diagnosis of schizoaffective disorder, bipolar disorder, depression with psychotic symptoms, or organic brain syndromes
* Meeting DSM-IV-TR criteria for any significant Psychoactive Substance Use Disorder within the 3 months prior to Screening
* Treatment-resistant to antipsychotic medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2005-06; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who discontinue because of Adverse Events

SECONDARY OUTCOMES:
Change in Clinical Global Impression scale, Investigator Assessment Questionnaire, cognitive functioning and outcome research assessments at endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (72):
- Austria (2):
  - Local Institution, Hall/Tirol
  - Local Institution, Vienna
- Belgium (6):
  - Local Institution, Bruges
  - Local Institution, Brussels
  - Local Institution, Diest
  - Local Institution, Halle
  - Local Institution, Sint-Denijs-Westrem
  - Local Institution, Stokrooie
- Czechia (4):
  - Local Institution, Havířov
  - Local Institution, Olomouc
  - Local Institution, Prague
  - Local Institution, Přerov
- France (16):
  - Local Institution, Aubagne
  - Local Institution, Bordeaux
  - Local Institution, Brumath
  - Local Institution, Château-Gontier
  - Local Institution, Clermont-Ferrand
  - Local Institution, Dijon
  - Local Institution, Dommartin-lès-Toul
  - Local Institution, Fains-Véel
  - Local Institution, Hénin-Beaumont
  - Local Institution, Le Pecq
  - Local Institution, Lyon
  - Local Institution, Poitiers
  - Local Institution, Reims
  - Local Institution, Roubaix
  - Local Institution, Toulon
  - Local Institution, Toulouse
- Germany (9):
  - Local Institution, Achim
  - Local Institution, Bochum
  - Local Institution, Cologne
  - Local Institution, Ellwangen
  - Local Institution, Hattingen
  - Local Institution, Neurnberg
  - Local Institution, Osnabrück
  - Local Institution, Ostfildern
  - Local Institution, Witten
- Greece (6):
  - Local Institution, Athens
  - Local Institution, Chania-Crete
  - Local Institution, Corfu
  - Local Institution, Leros
  - Local Institution, Thessaloniki
  - Local Institution, Tripoli
- Hungary (6):
  - Local Institution, Baja
  - Local Institution, Eger
  - Local Institution, Esztergom
  - Local Institution, Kistarcsa
  - Local Institution, Pécs
  - Local Institution, Sopron
- Italy (8):
  - Local Institution, Sestri Ponente, Genova
  - Local Institution, Aosta
  - Local Institution, Bolzano
  - Local Institution, Foggia
  - Local Institution, L’Aquila
  - Local Institution, Milan
  - Local Institution, Roggiano Gravina (Cs)
  - Local Institution, Roma
- Spain (10):
  - Local Institution, Terrassa, Barcelona
  - Local Institution, Barcelona
  - Local Institution, Elche (Alicante)
  - Local Institution, Langreo-Asturias
  - Local Institution, Madrid
  - Local Institution, Murcia
  - Local Institution, Oviedo
  - Local Institution, Salamanca
  - Local Institution, Valencia
  - Local Institution, Zamora
- United Kingdom (5):
  - Local Institution, Newport, Gwent
  - Local Institution, South Wales, Mid Glamorgan
  - Local Institution, Hull, North Yorkshire
  - Local Institution, Dundee, Tayside
  - Local Institution, Haywards Health, West Sussex

REFERENCES:
- [Background] Ryckmans V, Kahn JP, Modell S, Werner C, McQuade RD, Kerselaers W, Lissens J, Sanchez R. Switching to aripiprazole in outpatients with schizophrenia experiencing insufficient efficacy and/or safety/tolerability issues with risperidone: a randomized, multicentre, open-label study. Pharmacopsychiatry. 2009 May;42(3):114-21. doi: 10.1055/s-0028-1112134. Epub 2009 May 18. PMID 19452380